CLINICAL TRIAL: NCT02458859
Title: A 100 Patient, Prospective, Randomised, Clinical Evaluation Comparing Clinical and Health Economic Outcomes Between Patients With Chronic or Sub-acute Wounds Treated With Either PICO or Standard Care Dressings and a Qualitative Study to Explore the Experiences of Patients Receiving PICO With Particular Emphasis on Concordance
Brief Title: Trial of PICO Versus Standard Care in Chronic and Sub-acute Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE/044/PIC; NCT01683344 (obsolete NCT alias)
Record Dates: First submitted 2011-08-18; First posted 2015-06-01 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Wounds
Keywords: Chronic; Subacute
MeSH Terms: conditions — Wounds and Injuries; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICO (Active Comparator): PICO Negative Pressure Wound Therapy (NPWT) system
  Interventions: Device: PICO (single use portable negative pressure wound therapy)
- Standard care (No Intervention): Standard care

INTERVENTIONS:
Device: PICO (single use portable negative pressure wound therapy) — Single use portable negative pressure wound therapy
  Arms: PICO

SUMMARY:
Randomised Controlled Trial of PICO (a portable Negative Pressure Wound Therapy) versus standard care in patients with chronic and sub-acute wounds. Sample size 100 patients to investigate Time to healing, health economic and patient reported outcomes.

DETAILED DESCRIPTION:
The current study is being conducted to assess the clinical and cost effectiveness of managing patients with a chronic or sub-acute wound in a community setting with PICO and to explore the patient experience and issues of concordance that affect patients treated with PICO. The study will provide information on the level of clinical benefit that PICO can deliver in the population studied in order to justify a sample size for a definitive evaluation of PICO and the study will further assess wound types that may benefit from treatment with PICO.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Males and females. If female, they must not be pregnant or lactating. If female and of reproductive age, a pregnancy test will be provided.
* The patient or their legal representative (if the patient is incapable of giving legal consent), is able to understand the trial and is willing to consent to the trial.
* Patients with sub-acute or chronic wounds (diabetic foot ulcer, pressure ulcer, venous leg ulcer, or other chronic) suitable for treatment with a PICO dressing.
* Wound duration ≤52 weeks - Amended to remove criteria.
* Wound area range ≥5 cm2 at start of screening period
* Wound maximum linear dimension ≤ 15cm
* Able to use English for the interview

Exclusion Criteria:

* Patients with known allergies to product components (silicone adhesives and polyurethane films (direct contact with wound), acrylic adhesives (direct contact with skin), polyethylene fabrics and super-absorbent powders (polyacrylates) (within the dressing).
* Wounds which have an infection which is not being treated with systemic antibiotics.
* Wounds which are actively bleeding.
* Exposure of blood vessels, organs, bone or tendon at the base of the reference wound
* Exclude undermining or tunnelling present or suspected in the wound
* Use of negative pressure device on wound in the last 30 days. Amended to remove criteria
* Malignant wounds/malignancy in the wound
* Systemic infection not being treated with systemic antibiotics
* Simultaneous treatment with other experimental wound care procedures, biologics or devices
* Patients with a known history of poor compliance with medical treatment.
* Patients who have participated in this trial previously and who closed or were withdrawn.
* Patients who are unable to understand the aims and objectives of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Time to closure | 12 weeks
  Time to complete wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Christine Moffatt, Prof, Principal Investigator — Royal Derby Hospitals NHS Foundation trust/Nottingham University
Locations (20):
- Nursing Practise Solutions, Altario, Canada
- United Kingdom (19):
  - Bradford District Care Trust, Bradford
  - Papworth Surgery, Cambridge
  - Cossington House Surgery, Canterbury
  - Richmond House Surgery, Crook of Devon
  - Barton Surgery, Dawlish
  - Derby Hospit6al NHS Foundation Trust, Derby
  - South Axholme Practice, Doncaster
  - Sea Road Surgery, Garway
  - Dr Moss & Partners, Harrogate
  - The Honiton Group Practise, Honiton
  - Leodis Care Limited, Leeds
  - Barlow Medical centre, Manchester
  - Wellfield Medical Centrre, Manchester
  - Southbourne Surgery, Milton of Campsie
  - Kiltearn Medical Centre, Nantwich
  - Northumbria Healthcare NHS Trust, Newcastle
  - South Tyneside NHS Foundation Trust, Newcastle
  - Dr Jones & Partners, Sedgefield
  - Brunel Medical practise, Torquay